CLINICAL TRIAL: NCT00722358
Title: Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Antiviral Activity and Safety, Tolerability, and Pharmacokinetics of BMS-650032 in Subjects Infected With Hepatitis C Virus Genotype 1
Brief Title: A Multiple Ascending Dose Study of BMS-650032 in HCV Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI447-004
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — asunaprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-650032 (Active Comparator)
  Interventions: Drug: BMS-650032
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-650032 — Capsule, Oral, Q12h, 3/5 days
  Panel 1: 200 mg
  Panel 2: 400 mg
  Panel 3: 600 mg
  Arms: BMS-650032
Drug: Placebo — Capsule, Oral, Q 12h, 3/5 days
  Panel 1: matching placebo
  Panel 2: matching placebo
  Panel 3: matching placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the change in HCV RNA during dosing with BMS-650032 and during the follow-up period in subjects with chronic hepatitis C infection

ELIGIBILITY:
Inclusion Criteria:

* Chronically infected with HCV genotype 1
* Treatment naive
* HCV RNA viral load of ≥10*5 IU/mL
* BMI 18 to 35kg/m²

Exclusion Criteria:

* Women of childbearing potential (WOCBP)
* Any significant acute or chronic medical illness which is not stable or is not controlled with medication and not consistent with HCV infection
* HCV infected subjects who are treatment non-responder (defined as subject who received at least 12 weeks of SOC and continue to have a detectable HCV RNA level or subjects who did not attain a 2-log decline in HCV RNA levels at 12 weeks and stopped treatment
* HCV infected subjects who are treatment intolerant (defined as subject who are unable to receive at least 12 weeks of SOC due to toxicities associated with interferon and/or ribavirin
* HIV and/or HBV positive
* Major surgery within 4 weeks of study drug administration and any gastrointestinal surgery that could impact the absorption of study drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Antiviral activity will be assessed by the magnitude and rate of change in plasma HCV RNA levels from baseline. The primary endpoint for antiviral activity is decrease from baseline in plasma HCV RNA levels to Day 3/ or 5 | To assess the change in HCV RNA during dosing with BMS-650032 from baseline to Day 3 and during follow-up period

SECONDARY OUTCOMES:
PD-PK Relationship Measures: Asses relationship between antiviral activity and measures of exposure to BMS-650032 | 28 days after drug
Safety Outcome Measures: Safety and tolerability assessments | will be performed for a period of 28 days after administration of multiple doses of BMS-650032 for 3/ or 5 days
Pharmacokinetic Measures: Pharmacokinetic assessments | will be done on Day 1 for one dosing interval after the AM dose and on Day 3/ or 5 for 72 hours after the last AM dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (4):
  - Advanced Clinical Res Inst, Anaheim, California
  - Orlando Clinical Research Center, Orlando, Florida
  - Parexel International Corporation, Baltimore, Maryland
  - Central Texas Clinical Research, Austin, Texas
- Local Institution, Santurce, Puerto Rico

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx